CLINICAL TRIAL: NCT05057468
Title: Cyclosporine As a Second-line Treatment of Primary Autoimmune Hemolytic Anemia
Brief Title: Second-line Treatment of Primary Autoimmune Hemolytic Anemia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ghada E. M. Abdallah, lecturer in internal medicine department of faculty of medicine,Assiut university, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17300534
Record Dates: First submitted 2021-09-16; First posted 2021-09-27 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Primary Autoimmune Hemolytic Anemia
MeSH Terms: interventions — Cyclosporine; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cyclosporine (Experimental): 2.5-5mg/kg of cyclosporine daily for 3 months
  Interventions: Drug: Cyclosporine
- Rituximab (Active Comparator): 375 mg/ m2 weekly dose for a maximum of 4 weeks.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Cyclosporine — 2.5-5 mg orally for 3 months
  Arms: Cyclosporine
Drug: Rituximab — 375 mg/ m2 weekly dose for a maximum of 4 weeks
  Arms: Rituximab

SUMMARY:
the cyclosporine showed efficacy in many immune cytopenic diseases in the light of numerous case reports and retrospective data. This study compares cyclosporin versus rituximab in steroid-refractory anemia.

DETAILED DESCRIPTION:
Auto-immune hemolytic anemia (AIHA) is a heterogeneous syndrome in adults. This disease is associated with significant morbidity-mortality. First-line treatment with prolonged corticosteroid is well identified but there is not enough data about cyclosporine treatment in case of resistance or dependence on steroids.

the cyclosporine showed efficacy in many immune cytopenic diseases in the light of numerous case reports and retrospective data. This drug is cheap, licensed in immunologic diseases, and does not expose to major infections. So, we compare cyclosporin versus rituximab in steroid-refractory anemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged more than 18 years old from any sex with a diagnosis of primary warm autoimmune hemolytic anemia (AIHA) based on the presence of hemolytic anemia and serological evidence of anti-erythrocyte antibodies, detectable by the direct antiglobulin test who have disease progression or failure after treatment with steroid therapy, or who are intolerant to treatment, or who refuse standard treatment.
* No evidence of a lymphoproliferative malignancy or other autoimmune-related underlying conditions.

Exclusion Criteria:

* any contraindications to the drugs of the study.
* any identified secondary cause of the AIHA.
* pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-10-20 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
the proportion of complete response | 3months
  Hb ≥12 g/dL and normalization of all hemolytic markers
the proportion of partial response | 3months
  (Hb ≥10 g/dL or at least 2 g/dL increase in Hb, and no transfusion requirement

SECONDARY OUTCOMES:
rate of adverse events | 3months
  according to Common Terminology Criteria for Adverse Events Version 5

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university hospital, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No